CLINICAL TRIAL: NCT03330106
Title: A Randomized, Crossover Phase 1 Study to Evaluate the Effects of Pevonedistat on the QTc Interval in Patients With Advanced Solid Tumors
Brief Title: A Study to Evaluate the Effects of Pevonedistat on the Corrected QT (QTc) Interval in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Pevonedistat-1014; 2017-002610-31 (EudraCT Number); U1111-1201-10111 (Registry Identifier: WHO)
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Results first posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2022-06

CONDITIONS: Advanced Solid Neoplasm
Keywords: Drug therapy
MeSH Terms: interventions — pevonedistat; Docetaxel; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: Pevonedistat 25 mg/m^2 + Pevonedistat 50 mg/m^2 (Experimental): Pevonedistat 25 mg/m^2, infusion, intravenously, once on Day 1 of Cycle 1, followed by pevonedistat 50 mg/m^2, infusion, intravenously, once on Day 8 of Cycle 1.
  Interventions: Drug: Pevonedistat
- Part A: Pevonedistat 50 mg/m^2 + Pevonedistat 25 mg/m^2 (Experimental): Pevonedistat 50 mg/m^2, infusion, intravenously, once on Day 1 of Cycle 1, followed by pevonedistat 25 mg/m^2, infusion, intravenously, once on Day 8 of Cycle 1.
  Interventions: Drug: Pevonedistat
- Part B: Pevonedistat (Experimental): Pevonedistat 25 mg/m^2 in combination with docetaxel 75 mg/m^2 or pevonedistat 20 mg/m^2 in combination with carboplatin plus paclitaxel 175 mg/m^2, infusion, intravenously, once on Day 1 in each 21-day treatment cycle followed by pevonedistat 25 mg/m^2 or 20 mg/m^2 infusion, intravenously, once on Days 3 and 5 in each 21-day treatment cycle for up to 12 cycles or symptomatic deterioration or PD, treatment is discontinued for another reason, or until the study is stopped. The combination and dose of pevonedistat will be based on investigator discretion.
  Interventions: Drug: Pevonedistat; Drug: Docetaxel; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Pevonedistat — Pevonedistat intravenous infusion.
  Other Names: MLN4924, TAK-924
Drug: Docetaxel — Docetaxel intravenous infusion.
  Arms: Part B: Pevonedistat
Drug: Carboplatin — Carboplatin intravenous infusion.
  Arms: Part B: Pevonedistat
Drug: Paclitaxel — Paclitaxel intravenous infusion.
  Arms: Part B: Pevonedistat

SUMMARY:
The purpose of this study is to characterize the effects of 25 and 50 milligram per square meter (mg/m^2) pevonedistat on the Fridericia corrected QT interval (QTcF) of the electrocardiogram (ECG).

DETAILED DESCRIPTION:
The drug being tested in this study is called pevonedistat. Pevonedistat in combination with standard of care will be used to treat participants who have advanced solid tumors. This study will assess the effects of pevonedistat on the QTc interval in participants with advanced solid tumors.

The study will enroll approximately 45 participants. The study will be conducted in two Parts: Part A and Part B. Part A will have a 2-way crossover design and will involve the collection of triplicate ECGs. In Part A, participants will be randomly assigned to one of the two treatment groups as follow:

* Pevonedistat 25 mg/m^2 + Pevonedistat 50 mg/m^2
* Pevonedistat 50 mg/m^2 + Pevonedistat 25 mg/m^2

Eligible participants from Part A will continue treatment in optional Part B with pevonedistat in combination with SoC, docetaxel or carboplatin plus paclitaxel. The investigator will decide which pevonedistat combination a participant will receive.

* Pevonedistat 25 mg/m^2 + Docetaxel
* Pevonedistat 20 mg/m^2 + Carboplatin + Paclitaxel

This multi-center trial will be conducted in the United States. The overall time to participate in this study is 9.6 months. Participants will make a final visit to the clinic 30 days after receiving their last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have a histologically or cytologically confirmed metastatic or locally advanced solid tumor(s) appropriate for treatment with one of the 2 combination therapies in Part B of this study, have progressed despite standard therapy, or for whom conventional therapy is not considered effective.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
3. Expected survival longer than 3 months from enrollment in the study.
4. Recovered (that is, grade less than or equal to [<=] 1 toxicity) from the reversible effects of prior anticancer therapy.
5. Suitable venous access for the study-required blood sampling (including pharmacokinetic [PK] sampling).

Exclusion Criteria:

1. Treatment with strong cytochrome P3A (CYP3A) inducers within 14 days before the first dose of pevonedistat. Participants must have no history of amiodarone use within 6 months before the first dose of pevonedistat nor require the use of these medications during the study.
2. Treatment with QT-prolonging drugs with a risk of causing torsades de pointes (TdP. Participants taking drugs with a possible or conditional risk of QT prolongation or drugs that are to be avoided by participants with congenital long QT syndrome may be considered if on a stable dose, pending discussion and agreement between the investigator and the sponsor.
3. History of Brugada syndrome, risk factors for TdP, or family history of long QT syndrome.
4. Implantable cardioverter defibrillator.
5. Cardiac pacemaker with heart rate (HR) set at a fixed rate and treatment with concomitant medication that may limit increase in HR in response to hypotension (example, high-dose beta blocker).
6. Known moderate to severe aortic stenosis, moderate to severe mitral stenosis, or other valvulopathy (ongoing).
7. Admission or evidence of illicit drug use, drug abuse, or alcohol abuse.

Entry Criteria for Continuation to Optional Part B:

After completing Part A of the study, participants may choose to enter the optional Part B of the study. To be eligible for the optional Part B, participants must have completed Part A and be reassessed to determine if they meet the entry criteria for optional Part B. Only participants who meet the following criteria may enter into Part B:

* ECOG performance status of 0 to 1.
* Absolute neutrophil count (ANC) greater than or equal to (>=) 1500 per cubic millimeter (/mm^3).
* Platelet count >=100,000/mm^3.
* Laboratory values for hemoglobin, total bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), and serum creatinine or calculated/measured creatinine clearance.
* Diarrhea symptoms resolved to Grade 1 or better.
* QTc interval <480 millisecond (msec).
* Computed tomography (CT) scan or magnetic resonance imaging (MRI) of the chest, abdomen, and pelvis within 28 days of Cycle 1 Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2021-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (8):
- United States (8):
  - Sarcoma Oncology Center, Santa Monica, California
  - Moffitt Cancer Center, Tampa, Florida
  - Henry Ford Hospital, Detroit, Michigan
  - Montefiore Medical Center, The Bronx, New York
  - Case Western Reserve University, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mary Crowley Medical Research, Dallas, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Zhou X, Richardson DL, Dowlati A, Goel S, Sahebjam S, Strauss J, Chawla S, Wang D, Mould DR, Samnotra V, Faller DV, Venkatakrishnan K, Gupta N. Effect of Pevonedistat, an Investigational NEDD8-Activating Enzyme Inhibitor, on the QTc Interval in Patients With Advanced Solid Tumors. Clin Pharmacol Drug Dev. 2023 Mar;12(3):257-266. doi: 10.1002/cpdd.1194. Epub 2022 Nov 16. PMID 36382849

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 44 participants took part in this study at 8 investigative sites in the United States from 15 November 2017 to 21 June 2021.
Pre-assignment Details: Participants with histologically or cytologically confirmed metastatic or locally advanced solid tumor were enrolled in this 2-part study to receive intravenous infusion of pevonedistat in Part A and pevonedistat in combination with chemotherapy agents in Part B (optional part). After completion of Part A, participants had an opportunity to continue into optional Part B.
Groups:
- Part A: Pevonedistat 25 mg/m^2 + Pevonedistat 50 mg/m^2: Pevonedistat 25 mg/m^2, infusion, intravenously (IV), once on Day 1, followed by pevonedistat 50 mg/m^2, infusion, IV, once on Day 8 in Part A.
- Part A: Pevonedistat 50 mg/m^2 + Pevonedistat 25 mg/m^2: Pevonedistat 50 mg/m^2, infusion, IV, once on Day 1, followed by pevonedistat 25 mg/m^2, infusion, IV, once on Day 8 in Part A.
- Part B: Pevonedistat 25 mg/m^2 + Docetaxel: Pevonedistat 25 mg/m^2 in combination with docetaxel 75 mg/m^2, infusion, IV, once on Day 1 followed by pevonedistat 25 mg/m^2 IV, once on Days 3 and 5 in each 21-day treatment cycle for up to Cycle 45 or symptomatic deterioration or progressive disease (PD), or until treatment is discontinued for another reason. Pevonedistat was administered after the docetaxel chemotherapy. Participants who completed Part A and provided consent for Part B continued treatment in Part B.
- Part B: Pevonedistat 20 mg/m^2 + Carboplatin + Paclitaxel: Pevonedistat 20 mg/m^2 in combination with carboplatin area under the plasma concentration (AUC) at the dose of 5 milligram per minute per milliliter (mg/min/mL), infusion, IV and paclitaxel 175 mg/m^2, infusion, IV, once on Day 1 in each 21-day treatment cycle followed by pevonedistat 20 mg/m^2 IV, once on Days 3 and 5 in each 21-day treatment cycle for up to 20 cycles or symptomatic deterioration or PD, or until treatment is discontinued for another reason. Pevonedistat was administered after the paclitaxel and carboplatin chemotherapy. Participants who completed Part A and provided consent for Part B continued treatment in Part B.
Period: Part A
Arm/Group | Part A: Pevonedistat 25 mg/m^2 + Pevonedistat 50 mg/m^2 | Part A: Pevonedistat 50 mg/m^2 + Pevonedistat 25 mg/m^2 | Part B: Pevonedistat 25 mg/m^2 + Docetaxel | Part B: Pevonedistat 20 mg/m^2 + Carboplatin + Paclitaxel
Started | 22 | 22 | 0 | 0
Completed | 18 | 17 | 0 | 0
Not Completed | 4 | 5 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Death | 2 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Subjects Outside Eligibility Window for Part B due to Serious Adverse Event (SAE) | 0 | 1 | 0 | 0
Not completed — Worsening Creatinine Clearance and Thrombocytopenia | 1 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 1 | 0 | 0
Period: Part B
Arm/Group | Part A: Pevonedistat 25 mg/m^2 + Pevonedistat 50 mg/m^2 | Part A: Pevonedistat 50 mg/m^2 + Pevonedistat 25 mg/m^2 | Part B: Pevonedistat 25 mg/m^2 + Docetaxel | Part B: Pevonedistat 20 mg/m^2 + Carboplatin + Paclitaxel
Started (Participants who completed Part A were randomized in Part B to receive pevonedistat in combination with standard of care agents, either docetaxel or carboplatin+paclitaxel, as recommended by the Investigator.) | 0 | 0 | 23 | 12
Completed | 0 | 0 | 5 | 4
Not Completed | 0 | 0 | 18 | 8
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 0
Not completed — Death | 0 | 0 | 2 | 0
Not completed — Clinical Progression | 0 | 0 | 1 | 1
Not completed — Symptomatic Deterioration | 0 | 0 | 0 | 1
Not completed — Symptomatic Deterioration, Participant Placed on Hospice | 0 | 0 | 0 | 1
Not completed — Progressive Disease | 0 | 0 | 11 | 4

BASELINE CHARACTERISTICS:
Population: Randomized Population included all participants who had a randomization date and had been randomized to a treatment sequence.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Pevonedistat 25 mg/m^2 + Pevonedistat 50 mg/m^2 | Part A: Pevonedistat 50 mg/m^2 + Pevonedistat 25 mg/m^2 | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (9.15) | 59.5 (11.36) | 60.3 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 18 | 31
  Male | 9 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 17 | 18 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 16 | 17 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Part A: Change From Time-matched Baseline in Fridericia-corrected QT Interval (QTcF) After Pevonedistat Administration
Description: Change from time-matched baseline in QTcF was assessed following a single intravenous dose administration of pevonedistat at 25 and 50 mg/m^2 and was analysed by dose. Some participants were treated with pevonedistat 25 mg/m^2 or 50 mg/m^2 on Day 1 while others received treatment on Day 8. Data is reported at pre-dose and at multiple timepoints (1, 2, 3, 4, 6, 9, 11 and 24 hours) postdose up to Day 8 in Part A. Analysis of variance (ANOVA) was used for the analysis.
Time Frame: Baseline up to Day 8
Population: QT Population included all participants who received the protocol-specified pevonedistat dosing and had sufficient electrocardiogram (ECG) assessments in the Baseline period (Day -1) and at least one period of assessment of effect of pevonedistat (Day 1 or Day 8) to permit reliable analysis. Overall number analyzed are the number of participants with evaluable data for analyses by dose. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Groups:
- Pevonedistat 25 mg/m^2: Pevonedistat 25 mg/m^2, infusion, IV, once on Day 1 or Day 8.
- Pevonedistat 50 mg/m^2: Pevonedistat 50 mg/m^2, infusion, IV, once on Day 1 or Day 8.
Arm/Group | Pevonedistat 25 mg/m^2 | Pevonedistat 50 mg/m^2
Number analyzed (Participants) | 42 | 40
milliseconds
  Predose: number analyzed (Participants) | 41 | 40
  Predose | 1.310 [-2.238 to 4.857] | -2.231 [-5.790 to 1.328]
  1 Hour Postdose: number analyzed (Participants) | 41 | 39
  1 Hour Postdose | 3.180 [-0.367 to 6.727] | -0.639 [-4.213 to 2.935]
  2 Hours Postdose | 0.840 [-2.694 to 4.375] | -2.127 [-5.688 to 1.434]
  3 Hours Postdose | 1.754 [-1.783 to 5.291] | -1.184 [-4.747 to 2.379]
  4 Hours Postdose: number analyzed (Participants) | 41 | 40
  4 Hours Postdose | 2.567 [-0.980 to 6.114] | -1.127 [-4.688 to 2.434]
  6 Hours Postdose: number analyzed (Participants) | 40 | 39
  6 Hours Postdose | 0.598 [-2.963 to 4.159] | -3.465 [-7.040 to 0.111]
  9 Hours Postdose: number analyzed (Participants) | 41 | 39
  9 Hours Postdose | -2.998 [-6.548 to 0.552] | -6.898 [-10.475 to -3.322]
  11 Hours Postdose: number analyzed (Participants) | 35 | 32
  11 Hours Postdose | -2.478 [-6.113 to 1.158] | -8.638 [-12.330 to -4.946]
  24 Hours Postdose: number analyzed (Participants) | 35 | 34
  24 Hours Postdose | -2.930 [-6.566 to 0.706] | -7.653 [-11.307 to -4.000]

2. Secondary Outcome: Part A: Change From Time-matched Baseline in Individual Corrected QT Interval (QTcI) After Pevonedistat Administration
Description: Change from time-matched baseline in QTcI was assessed following a single intravenous dose administration of pevonedistat at 25 and 50 mg/m^2 and was analysed by dose. Some participants were treated with pevonedistat 25 mg/m^2 or 50 mg/m^2 on Day 1 while others received treatment on Day 8. ANOVA was used for the analysis.
Time Frame: Predose, and at multiple time points up to 24 hours post dose on Day 1 or Day 8 in Part A
Population: QT Population included all participants who received the protocol-specified pevonedistat dosing and had sufficient ECG assessments in the Baseline period (Day -1) and at least one period of assessment of effect of pevonedistat (Day 1 or Day 8) to permit reliable analysis. Overall number analyzed are the number of participants with evaluable data for analyses by dose. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Arm/Group | Pevonedistat 25 mg/m^2 | Pevonedistat 50 mg/m^2
Number analyzed (Participants) | 42 | 40
milliseconds
  Predose: number analyzed (Participants) | 41 | 40
  Predose | 2.099 [-2.860 to 7.058] | -1.884 [-6.852 to 3.084]
  1 Hour Postdose: number analyzed (Participants) | 41 | 39
  1 Hour Postdose | 3.580 [-1.378 to 8.538] | -0.206 [-5.185 to 4.774]
  2 Hours Postdose | 1.477 [-3.471 to 6.425] | -0.099 [-5.068 to 4.870]
  3 Hours Postdose | 3.074 [-1.877 to 8.024] | 1.877 [-3.093 to 6.848]
  4 Hours Postdose: number analyzed (Participants) | 41 | 40
  4 Hours Postdose | 3.816 [-1.144 to 8.776] | 1.305 [-3.665 to 6.275]
  6 Hours Postdose: number analyzed (Participants) | 40 | 39
  6 Hours Postdose | 2.143 [-2.826 to 7.112] | 0.198 [-4.783 to 5.179]
  9 Hours Postdose: number analyzed (Participants) | 41 | 39
  9 Hours Postdose | -1.419 [-6.378 to 3.540] | -2.482 [-7.462 to 2.499]
  11 Hours Postdose: number analyzed (Participants) | 35 | 32
  11 Hours Postdose | 0.020 [-5.009 to 5.049] | -5.250 [-10.323 to -0.177]
  24 Hours Postdose: number analyzed (Participants) | 35 | 34
  24 Hours Postdose | -1.897 [-6.926 to 3.132] | -3.105 [-8.147 to 1.937]

3. Secondary Outcome: Part A: Change From Time-matched Baseline in QRS After Pevonedistat Administration
Description: Change from time-matched baseline in QRS was assessed following a single intravenous dose administration of pevonedistat at 25 and 50 mg/m^2 and was analysed by dose. Some participants were treated with pevonedistat 25 mg/m^2 or 50 mg/m^2 on Day 1 while others received treatment on Day 8. ANOVA was used for the analysis.
Time Frame: Predose, and at multiple time points post dose up to 24 hours on Day 1 or Day 8 in Part A
Population: as for outcome 2
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Arm/Group | Pevonedistat 25 mg/m^2 | Pevonedistat 50 mg/m^2
Number analyzed (Participants) | 42 | 40
milliseconds
  Predose: number analyzed (Participants) | 41 | 40
  Predose | -0.459 [-2.687 to 1.768] | -0.482 [-2.713 to 1.748]
  1 Hour Postdose: number analyzed (Participants) | 41 | 39
  1 Hour Postdose | 1.447 [-0.780 to 3.675] | 0.850 [-1.384 to 3.084]
  2 Hours Postdose | -0.212 [-2.437 to 2.013] | -0.043 [-2.274 to 2.188]
  3 Hours Postdose | 0.138 [-2.088 to 2.363] | 0.184 [-2.048 to 2.415]
  4 Hours Postdose: number analyzed (Participants) | 41 | 40
  4 Hours Postdose | -1.068 [-3.296 to 1.159] | -0.241 [-2.471 to 1.990]
  6 Hours Postdose: number analyzed (Participants) | 40 | 39
  6 Hours Postdose | -0.192 [-2.423 to 2.038] | -0.319 [-2.552 to 1.915]
  9 Hours Postdose: number analyzed (Participants) | 41 | 39
  9 Hours Postdose | -0.791 [-3.019 to 1.437] | -0.221 [-2.455 to 2.013]
  11 Hours Postdose: number analyzed (Participants) | 35 | 32
  11 Hours Postdose | -0.551 [-2.799 to 1.696] | -0.769 [-3.029 to 1.491]
  24 Hours Postdose: number analyzed (Participants) | 35 | 34
  24 Hours Postdose | -0.946 [-3.193 to 1.301] | -0.470 [-2.721 to 1.781]

4. Secondary Outcome: Part A: Change From Time-matched Baseline in PR After Pevonedistat Administration
Description: Change from time-matched baseline in PR was assessed following a single intravenous dose administration of pevonedistat at 25 and 50 mg/m^2 and was analysed by dose. Some participants were treated with pevonedistat 25 mg/m^2 or 50 mg/m^2 on Day 1 while others received treatment on Day 8. ANOVA was used for the analysis.
Time Frame: Predose, and at multiple time points post dose up to 24 hours on Day 1 or Day 8 in Part A
Population: as for outcome 2
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Arm/Group | Pevonedistat 25 mg/m^2 | Pevonedistat 50 mg/m^2
Number analyzed (Participants) | 42 | 40
milliseconds
  Predose: number analyzed (Participants) | 41 | 39
  Predose | -2.894 [-8.227 to 2.440] | -1.220 [-6.563 to 4.122]
  1 Hour Postdose: number analyzed (Participants) | 41 | 38
  1 Hour Postdose | 1.152 [-4.181 to 6.486] | 3.360 [-1.989 to 8.709]
  2 Hours Postdose: number analyzed (Participants) | 42 | 39
  2 Hours Postdose | -0.090 [-5.419 to 5.240] | 1.514 [-3.830 to 6.857]
  3 Hours Postdose: number analyzed (Participants) | 42 | 39
  3 Hours Postdose | -1.557 [-6.886 to 3.773] | -0.167 [-5.510 to 5.177]
  4 Hours Postdose: number analyzed (Participants) | 41 | 39
  4 Hours Postdose | -3.406 [-8.740 to 1.927] | -1.802 [-7.146 to 3.542]
  6 Hours Postdose: number analyzed (Participants) | 40 | 38
  6 Hours Postdose | -4.665 [-10.004 to 0.674] | -4.463 [-9.812 to 0.887]
  9 Hours Postdose: number analyzed (Participants) | 41 | 38
  9 Hours Postdose | -4.499 [-9.833 to 0.836] | -3.608 [-8.957 to 1.742]
  11 Hours Postdose: number analyzed (Participants) | 35 | 31
  11 Hours Postdose | -3.018 [-8.385 to 2.349] | -2.333 [-7.729 to 3.062]
  24 Hours Postdose: number analyzed (Participants) | 34 | 33
  24 Hours Postdose | -5.245 [-10.617 to 0.128] | -6.499 [-11.878 to -1.120]

5. Secondary Outcome: Part A: Change From Time-matched Baseline in Heart Rate (HR) After Pevonedistat Administration
Description: Change from time-matched baseline in HR was assessed following a single intravenous dose administration of pevonedistat at 25 and 50 mg/m^2 and was analysed by dose. Some participants were treated with pevonedistat 25 mg/m^2 or 50 mg/m^2 on Day 1 while others received treatment on Day 8. ANOVA was used for the analysis.
Time Frame: Predose, and at multiple time points post dose up to 24 hours on Day 1 or Day 8 in Part A
Population: as for outcome 2
Measure: Least Squares Mean (90% Confidence Interval); unit: beats per minute (bpm)
Arm/Group | Pevonedistat 25 mg/m^2 | Pevonedistat 50 mg/m^2
Number analyzed (Participants) | 42 | 40
beats per minute (bpm)
  Predose: number analyzed (Participants) | 41 | 40
  Predose | 0.602 [-2.627 to 3.831] | 0.981 [-2.258 to 4.220]
  1 Hour Postdose: number analyzed (Participants) | 41 | 39
  1 Hour Postdose | -2.068 [-5.297 to 1.162] | -1.595 [-4.848 to 1.659]
  2 Hours Postdose | -1.812 [-5.030 to 1.406] | -0.556 [-3.797 to 2.686]
  3 Hours Postdose | -0.993 [-4.212 to 2.225] | 1.929 [-1.313 to 5.171]
  4 Hours Postdose: number analyzed (Participants) | 41 | 40
  4 Hours Postdose | -0.279 [-3.507 to 2.950] | 2.736 [-0.504 to 5.977]
  6 Hours Postdose: number analyzed (Participants) | 40 | 39
  6 Hours Postdose | 2.712 [-0.536 to 5.960] | 6.411 [3.150 to 9.671]
  9 Hours Postdose: number analyzed (Participants) | 41 | 39
  9 Hours Postdose | 2.545 [-0.686 to 5.775] | 7.134 [3.879 to 10.389]
  11 Hours Postdose: number analyzed (Participants) | 35 | 32
  11 Hours Postdose | 2.794 [-0.517 to 6.105] | 7.511 [4.149 to 10.872]
  24 Hours Postdose: number analyzed (Participants) | 35 | 34
  24 Hours Postdose | 4.432 [1.124 to 7.740] | 7.609 [4.288 to 10.930]

6. Secondary Outcome: Part A: Cmax: Maximum Observed Plasma Concentration for Pevonedistat
Time Frame: Days 1 or 8 predose and at multiple time points (up to 24 hours) post dose in Part A
Population: Pharmacokinetic (PK) Population included all participants who received the protocol-specified pevonedistat dosing during Part A and had sufficient PK assessments to permit reliable estimation of PK parameters. Overall number analyzed are the number of participants with evaluable data for analyses by dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Pevonedistat 25 mg/m^2 | Pevonedistat 50 mg/m^2
Number analyzed (Participants) | 44 | 43
nanograms per milliliter (ng/mL) | 197 (38.7) | 509 (35.6)

7. Secondary Outcome: Part A: AUC(0-24): Area Under the Plasma Concentration-time Curve From Time 0 to 24 Hours Postdose for Pevonedistat
Time Frame: Days 1 or 8 predose and at multiple time points (up to 24 hours) post dose in Part A
Population: PK Population included all participants who received the protocol-specified pevonedistat dosing during Part A and had sufficient PK assessments to permit reliable estimation of PK parameters. Overall number analyzed are the number of participants with evaluable data for analyses by dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Pevonedistat 25 mg/m^2 | Pevonedistat 50 mg/m^2
Number analyzed (Participants) | 43 | 43
hour*nanogram per milliliter (h*ng/mL) | 1190 (22.0) | 2510 (25.2)

8. Secondary Outcome: Part A: Terminal Phase Elimination Half-life (t1/2) for Pevonedistat
Time Frame: Days 1 or 8 predose and at multiple time points (up to 24 hours) post dose in Part A
Population: PK Population included all participants who received the protocol-specified pevonedistat dosing during Part A and had sufficient PK assessments to permit reliable estimation of PK parameters. Overall number analyzed are the number of participants with evaluable data for analyses.
Measure: Mean (Standard Deviation); unit: hours (h)
Arm/Group | Pevonedistat 25 mg/m^2 | Pevonedistat 50 mg/m^2
Number analyzed (Participants) | 43 | 42
hours (h) | 7.21 (1.35) | 6.73 (1.15)

9. Secondary Outcome: Part B: Overall Response Rate (ORR)
Description: Percentage of participants who achieve an overall response per investigator's assessment at end of treatment,according to Response Evaluation Criteria in Solid Tumor(RECIST),version 1.1 guideline. Complete response(CR):Disappearance of all target lesions.Any pathological lymph nodes(whether target and non target)must have reduction in short axis to <10 millimeter(mm).Partial Response(PR):atleast 30% decrease in sum of diameter of target lesions,taking as reference baseline sum of diameter.Stable Disease(SD):Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression(PD),taking as reference smallest sum of diameter; PD:atleast 20% increase in sum of diameter of target lesions,taking as reference,smallest sum on study(this includes baseline sum if that is smallest on study).In addition to relative increase of 20%,sum must also demonstrate an absolute increase of atleast 5 mm.Appearance of 1 or more new lesions is also considered progression.
Time Frame: Up to Cycle 45 (end of treatment) (Cycle length=21 days)
Population: Disease-response population included participants who received at least 1 dose of study drug in Part B, had measurable disease as entry criteria for Part B, and had at least 1 postbaseline disease assessment.
Measure: Number; unit: percentage of participants
Groups:
- Part B: Pevonedistat 20 mg/m^2 + Carboplatin + Paclitaxel: Pevonedistat 20 mg/m^2 in combination with carboplatin area under the plasma concentration (AUC) at the dose of 5 mg/min/mL, infusion, IV and paclitaxel 175 mg/m^2, infusion, IV, once on Day 1 in each 21-day treatment cycle followed by pevonedistat 20 mg/m^2 IV, once on Days 3 and 5 in each 21-day treatment cycle for up to 20 cycles or symptomatic deterioration or PD, or until treatment is discontinued for another reason. Pevonedistat was administered after the paclitaxel and carboplatin chemotherapy. Participants who completed Part A and provided consent for Part B continued treatment in Part B.
Arm/Group | Part B: Pevonedistat 25 mg/m^2 + Docetaxel | Part B: Pevonedistat 20 mg/m^2 + Carboplatin + Paclitaxel
Number analyzed (Participants) | 22 | 12
percentage of participants | 9.1 [1.0 to 10] | 8.3 [6.2 to 9.1]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to approximately 188 weeks (up to approximately 3.6 years)
Description: Safety Population for Part A included all participants who received at least 1 dose of pevonedistat during Part A. Safety population for Part B included all participants who continued to Part B and received at least 1 dose of study drugs during Part B. For Part A, MedDRA Version 22.0 was used and for Part B MedDRA version 24.0 was used.
Arm/Group | Part A: Pevonedistat 25 mg/m^2 + Pevonedistat 50 mg/m^2 | Part A: Pevonedistat 50 mg/m^2 + Pevonedistat 25 mg/m^2 | Part B: Pevonedistat 25 mg/m^2 + Docetaxel | Part B: Pevonedistat 20 mg/m^2 + Carboplatin + Paclitaxel
All-Cause Mortality (participants affected / at risk) | 2/22 | 4/22 | 2/23 | 0/12
Serious Adverse Events (participants affected / at risk) | 3/22 | 5/22 | 13/23 | 5/12
Other Adverse Events (participants affected / at risk) | 13/22 | 17/22 | 23/23 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Part A: Pevonedistat 25 mg/m^2 + Pevonedistat 50 mg/m^2 (N=22) | Part A: Pevonedistat 50 mg/m^2 + Pevonedistat 25 mg/m^2 (N=22) | Part B: Pevonedistat 25 mg/m^2 + Docetaxel (N=23) | Part B: Pevonedistat 20 mg/m^2 + Carboplatin + Paclitaxel (N=12)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Disseminated varicella zoster virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 0
Pyrexia (General disorders) | 0 | 0 | 2 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 2 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/13 | 0/18 | 1/16 | 0/7 — The number of participants exposed to this adverse event is based on the female population.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Pevonedistat 25 mg/m^2 + Pevonedistat 50 mg/m^2 (N=22) | Part A: Pevonedistat 50 mg/m^2 + Pevonedistat 25 mg/m^2 (N=22) | Part B: Pevonedistat 25 mg/m^2 + Docetaxel (N=23) | Part B: Pevonedistat 20 mg/m^2 + Carboplatin + Paclitaxel (N=12)
Aspartate aminotransferase increased (Investigations) | 4 | 3 | 7 | 5
Nausea (Gastrointestinal disorders) | 4 | 4 | 11 | 8
Alanine aminotransferase increased (Investigations) | 4 | 2 | 7 | 8
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 11 | 2
Fatigue (General disorders) | 2 | 3 | 17 | 10
Vomiting (Gastrointestinal disorders) | 0 | 4 | 5 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 4 | 3 | 5
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 8 | 4
Hypertension (Vascular disorders) | 0 | 3 | 5 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 9 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 7 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 6 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 3 | 1
Pyrexia (General disorders) | 2 | 0 | 4 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 5 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 6 | 5
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 2 | 3 | 1
Pain (General disorders) | 0 | 0 | 0 | 5
Oedema peripheral (General disorders) | 0 | 0 | 4 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 2
Chills (General disorders) | 0 | 0 | 3 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 3 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 3 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 6 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 4 | 5
Dysgeusia (Nervous system disorders) | 0 | 0 | 5 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 4
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 3
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 3
Syncope (Nervous system disorders) | 0 | 0 | 2 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 2
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 1
Drooling (Nervous system disorders) | 0 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 1
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 4 | 3
Neutrophil count decreased (Investigations) | 0 | 0 | 2 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 2 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 2 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 2
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1
Urine output decreased (Investigations) | 0 | 0 | 0 | 1
Vitamin D decreased (Investigations) | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 8 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 2 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 2 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 2
Incision site oedema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 2
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 2
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 2 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 2 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (2):
  • Study Protocol (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/06/NCT03330106/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/06/NCT03330106/SAP_001.pdf